CLINICAL TRIAL: NCT03538379
Title: Evaluation of Hemorrhage Control and Tourniquet Training Effectiveness for Laypersons
Brief Title: Tourniquet Training Effectiveness Study
Acronym: TRIAGE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: The Gillian Reny Stepping Strong Center for Trauma Innovation (Unknown)
Responsible Party: Principal Investigator, Eric Goralnick, Assistant Professor, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2018P000536
Record Dates: First submitted 2018-04-09; First posted 2018-05-29 (Actual); Last update posted 2018-05-29 (Actual); Status verified 2018-05

CONDITIONS: Trauma Injury; Hemorrhage
Keywords: Tourniquets; Bleeding Control Basic (B-Con) Course; Layperson training
MeSH Terms: conditions — Accidental Injuries; Hemorrhage

STUDY DESIGN:
Intervention Model Description: Individuals will complete the bleeding control basic (B-Con) course followed by evaluation of individuals ability to apply each of 5 different types of tourniquets. Each individual is evaluated for all 5 types of tourniquets. The order of testing for tourniquets for each individual is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Combat Application Tourniquet (CAT) (Active Comparator): The combat application tourniquet (CAT) is the type of commercial tourniquet taught in the B-Con course as administered by the investigators. It will serve as the control group to which all other types of tourniquets, which are not explicitly taught in the course, are compared to.
  Interventions: Behavioral: Bleeding Control Basic (B-Con) Course
- Sof Tourniquet (Sof-T) (Active Comparator): The Sof-Tourniquet (Sof-T) is a commercial windlass type tourniquet similar to the CAT tourniquet in that it is based on a windlass mechanism. Its application not explicitly taught in the B-Con course.
  Interventions: Behavioral: Bleeding Control Basic (B-Con) Course
- Stretch-Wrap-And-Tuck (SWAT) Tourniquet (Active Comparator): The Stretch-Wrap-And-Tuck (SWAT) Tourniquet is a commercial elastic tourniquet. Its application not explicitly taught in the B-Con course.
  Interventions: Behavioral: Bleeding Control Basic (B-Con) Course
- Rapid Application Tourniquet (RAT) (Active Comparator): The Rapid Application Tourniquet (RAT) is a commercial elastic tourniquet similar to a bungee cord. Its application not explicitly taught in the B-Con course.
  Interventions: Behavioral: Bleeding Control Basic (B-Con) Course
- Improvised Tourniquet (Active Comparator): The improvised tourniquet arm will involve participants being given supplies to enable them to fashion a tourniquet. The supplies will include a leather belt, gauze, shoestring, and a rod to act as a windlass.
  Interventions: Behavioral: Bleeding Control Basic (B-Con) Course

INTERVENTIONS:
Behavioral: Bleeding Control Basic (B-Con) Course — The American College of Surgeons Bleeding Control Basic Course will be provided to participants. This course consists of a 30-minute lecture followed by 30-minutes of hands-on training in hemorrhage control technique application. It teaches how to apply manual pressure and how to apply a Combat Application Tourniquet (CAT). The course will not vary from its typical administration for this study.

SUMMARY:
Trauma is the leading cause of death for individuals ages 1-45 years old, within this cohort, and uncontrolled hemorrhage is the leading cause of preventable death.1,2 Tourniquets have been shown to be effective in dramatically decreasing death from uncontrolled hemorrhage on the battlefield and there is level 4 evidence that EMS application of tourniquets in the civilian sector is effective though not to the same degree as in the military.3,4 Multiple national groups have advocated that to further decrease preventable deaths from hemorrhage, laypersons should apply tourniquets before the arrival of professional first responders. To this aim, the "Stop the Bleed" campaign has trained over 100,000 individuals in the US in hemorrhage control techniques and tourniquet use with the Bleeding Control Basic (B-Con) course.5 The "Stop the Bleed" campaign informs course participants all commercial tourniquets are equivalent, and improvised tourniquets should be applied if a commercial tourniquet is not available.6 The investigators are evaluating the ability of the B-Con course participants to apply three different types of commercial tourniquets, the Rapid Application tourniquet (RAT), the Stretch-Wrap-And-Tuck tourniquet (SWAT-T), and the Sof Tourniquet (Sof-T) as well as participants ability to fashion an improvised tourniquet. The investigators hypothesize B-Con in its current form does not enable course participants to apply other commercial tourniquets beyond the specific one taught, the CAT tourniquet, and does not teach how to apply an improvised tourniquet.

DETAILED DESCRIPTION:
Hemorrhage control by rapid application of commercial tourniquets has significantly improved the survival of military personnel injured on the battlefield.7,8 The U.S. civilian population has seen a spike in battlefield like injuries in the recent years, a prime example being the Boston Marathon bombing.9,10 To address this issue, the American College of Surgeons (ACS) formed a committee comprised of individuals from the fields of healthcare, law-enforcement, fire department, pre-hospital care and the military. This committee came up with a set of recommendation regarding first response and capacity building for hemorrhage control, known as the Harford Consensus.11 These recommendations include educational programs for lay-people in hemorrhage control with an emphasis on rapid and early tourniquet application. There is level 4 evidence that after adjustment for covariates, emergency medical providers' application of tourniquets in civilian trauma decreases mortality, though not to the same dramatic degree seen in the military setting.12-14 Researchers are working to show the effect of training of laypersons in hemorrhage control in the real world but no data beyond the simulation setting is currently presented in the literature.15 Various groups have developed training programs for hemorrhage control training, the most notable of which is the ACS "Stop the Bleed" Bleeding Control Basic (B-Con) training.16 B-Con has trained over 100,000 individuals in the US since its implementation.5 Goralnick et. al. have shown that there is moderate retention for the retention of B-Con specifically for application of the Combat Application Tourniquet (CAT), which is also the type of tourniquet with the best evidence for its use as it is the type used by the US military.17 However, the Hartford consensus and the "Stop the Bleed" campaign state that "(1) commercial windlass-type tourniquets should be used in the prehospital setting for the control of significant extremity hemorrhage when direct pressure is ineffective or impractical, (2) improvised tourniquets should be used only if no commercial device is available."5,18 This advocacy for types of commercial tourniquets beyond the CAT and, more significantly, for improvised tourniquets has not been studied in either a simulated or real setting.

There are multiple different tourniquet types available for which, while the principle is the same for all, the actual mechanism and steps for application vary. B-Con in its current iteration informs participants the principle is the same for both other commercial tourniquets and improvised tourniquets, which is to be tight enough to occlude arterial bleeding. Other courses which have been widely disseminated have taught how to use tourniquets other than the CAT, such as the Stretch-Wrap-And-Tuck tourniquet (SWAT-T).19 Currently, the courses being offered typically only teach how to use one, and sometimes two, different types of tourniquets. Furthermore, as there is not broad consensus statement about which tourniquet type to use and teach, different groups distribute different types of tourniquets in publicly available bleeding control kits, and professional first responders carry different types of commercial tourniquets. A randomized trial has shown that among some of the available commercial tourniquets, the CAT, ratcheting medical tourniquet (RMT), and SWAT-T, the proportion of application for those without training ranges from 10.6-23.4%.

The B-Con course presumption that participants understand tourniquet principles rather than a single technique, which would enable them to apply devices they have not seen before, has not been evaluated. In this context, the investigators would evaluate participants, immediately after completing the full B-Con course, on their ability to apply different commercial tourniquets than what they were trained on and their ability to apply a commercial tourniquet.

1. Study design:

   a) Prospective open-label trial
2. Consent:

   a) Verbal consent
3. Protocol:

   1. All participants will receive the ACS stop the Bleed training from qualified instructors. This training is 45 to 60 minutes long, consisting of an audio-visual presentation with tourniquet application instructions followed by hands-on training under the supervision of an instructor. The training takes place in groups of 20 to 50 at a time. The audio-visual part of the training takes place in groups of 20, which are then divided in to subgroups of 4-8 for hands-on training with an instructor. There is no compensation for the study participants.
   2. The evaluation of hemorrhage control competence will take place individually. A mannequin, the Hapmed tourniquet trainer, with a traumatic amputation of the leg just above the knee will be present. A reviewer will provide instructions, including that the lights on the leg represent continued bleeding and they will have a maximum of 2 minutes to apply the tourniquet. The participant will be provided a tourniquet and told to stop the simulated bleeding. Participants will be tested in all 5 types of tourniquets sequentially using the same method but with the order of testing varying according to the randomization. The reviewer will start timing after telling the participant to begin. This will then be repeated for the other type of tourniquet the individual will need to apply. No feedback will be given to the participant throughout the testing process.

   i) Supplies for the improvised tourniquet will include a T-shirt, long stretch of gauze, a stick to act as a windlass, and a leather belt c) Parameters measured: i) The participants will be timed until they feel that they have stopped the bleeding or they tell the instructor they are done. The maximum amount of time provided to apply the tourniquet will be 2 minutes based on the results of the investigators prior studies in which the 90th percentile for time to correct application was 117 seconds.

   ii) Appropriateness of hemorrhage control will be determined by correct placements of tourniquet as defined by at least 2 inches proximal to the amputation site iii) Adequate pressure to stop the bleeding which will be set at 250 mmHg. For unsuccessful hemorrhage control, the reason for failure will be recorded.

   iv) Correct tourniquet application defined by: (1) Time to application < 120 seconds (2) Placement of tourniquet a minimum of 2 inches proximal to amputation (3) Tourniquet application pressure > 250 mmHg d) All the reviewers would be physicians, nurses and EMTs, trained in hemorrhage-control. The complete test for each individual will not take more than 15 mins.
4. Randomization for the order of tourniquet application:

   a) Permutated block randomization will be used to vary the order for application of the 5 different types of tourniquets (CAT, RAT, SWAT-T, Sof-T, and improvised tourniquet)
5. Pre-trial questionnaire:

   a) Study subjects will be given a pre-trial questionnaire to gather information regarding age, gender, and level of education. The questionnaire will also include questions to assess their knowledge regarding hemorrhage control and to determine their willingness and self-reported comfort level in acting as a first-responder in a mass causality scenario. Answers will be presented on a Likert-type scale or dichotomous yes-no.
6. Post-trial questionnaire:

   a) After the hemorrhage control training, all participants will be given a questionnaire to evaluate comfort level, self-efficacy, and other questions relating to hemorrhage control response.
7. Sample size calculation:

   1. Sample Size calculation was done for paired comparisons with 80% power and Bonferroni corrected for 4 pairwise comparisons for an alpha level of 0.0125 and correlation of 0.1. The largest difference was then taken as the sample size for each arm.
   2. The expected corrected proportions for the different tourniquets are:

      1. CAT: 80-90% (Control)
      2. RAT: 10-30%
      3. SWAT-T: 10-30%
      4. Sof-T: 20-40%
      5. Improvised: < 10% ii) The smallest presumed difference in correct application for the CAT (control) at 80% is to the Sof-T at 40%. To attain 80% power with alpha of 0.0125 the required minimum sample size is 34.
   3. All sample size calculations performed using Stata v14.1.
8. Statistical Analysis:

   1. Paired statistical tests using McNemars test will be used for the univariate analysis of the primary outcome of correct tourniquet application comparing the CAT tourniquet as a control (CAT being type of tourniquet taught in the B-Con course) to each of the other tourniquet types (RAT, SWAT-T, Sof-T, Improvised) for 4 total pairwise comparisons.
   2. Descriptive statistical analysis (ANOVA, Kruskal-wallis, Mann Whitney U test, Student T-test) will be used to assess the secondary outcomes of time to tourniquet application, estimated blood loss prior to tourniquet application, and pressure applied by the tourniquet.
   3. Multiple Logistic regression will be used to assess for predictors of correct tourniquet application for each of the different tourniquet types. The model will include age, gender, education level, any prior hemorrhage control training, and success in application for each of the other tourniquet types.
   4. Descriptive statistics will also be used to assess participants responses on the questionnaires. Non-parametric statistical tests (Wilcoxon signed rank test and generalized estimating equations) will be used to assess 5-point Likert scale questions.
   5. P-value for significance will be set at 0.05 after Bonferroni correction.

ELIGIBILITY:
Inclusion Criteria:

* Participation in the Bleeding Control Basic Course

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2018-04-04 (Actual); Primary Completion 2018-06-30 (Estimated); Study Completion 2018-07-15 (Estimated)

PRIMARY OUTCOMES:
Correct Tourniquet Application | Within 30 minutes of completing training
  Correct tourniquet application for each type of tourniquet tested. Correct application for all arms / types of tourniquets is defined as application pressure > 250 mmHg, distance above injury of > 2 inches, and time to application < 2 minutes.

SECONDARY OUTCOMES:
Total Blood loss | Within 30 minutes of completing training
  Estimate of amount of blood loss prior to tourniquet application in milliliters.
Time to Tourniquet Application | Within 30 minutes of completing training
  Time to correct tourniquet application or participant stopping in seconds.
Pressure Applied by Tourniquet | Within 30 minutes of completing training
  Amount of pressure applied by the tourniquet measured in mmHg
Demographic Predictors of Correct Tourniquet Application | Within 30 minutes of completing training
  Demographics (age, gender, education level, prior training) associated with correct tourniquet application as defined as application pressure > 250 mmHg, distance above injury of > 2 inches, and time to application < 2 minutes.
Willingness-to-assist in Emergency | immediately before training and within 30 minutes of completing training
  Questions regarding willingness to assist in an emergency with responses reported on 5-point Likert Scale. 1 corresponds to very unwilling to assist and 5 corresponds to very willing to assist.
Comfort level Controlling Hemorrhage | immediately before training and within 30 minutes of completing training
  Questions regarding comfort level controlling hemorrhage with responses reported on 5-point Likert Scale. 1 corresponds to very uncomfortable and 5 corresponds to very comfortable controlling hemorrhage.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhee P, Joseph B, Pandit V, Aziz H, Vercruysse G, Kulvatunyou N, Friese RS. Increasing trauma deaths in the United States. Ann Surg. 2014 Jul;260(1):13-21. doi: 10.1097/SLA.0000000000000600. PMID 24651132
- [Background] Kwon AM, Garbett NC, Kloecker GH. Pooled preventable death rates in trauma patients : Meta analysis and systematic review since 1990. Eur J Trauma Emerg Surg. 2014 Jun;40(3):279-85. doi: 10.1007/s00068-013-0364-5. Epub 2014 Jan 29. PMID 26816061
- [Background] Kragh JF Jr, Walters TJ, Baer DG, Fox CJ, Wade CE, Salinas J, Holcomb JB. Survival with emergency tourniquet use to stop bleeding in major limb trauma. Ann Surg. 2009 Jan;249(1):1-7. doi: 10.1097/SLA.0b013e31818842ba. PMID 19106667
- [Background] Kauvar DS, Dubick MA, Walters TJ, Kragh JF Jr. Systematic review of prehospital tourniquet use in civilian limb trauma. J Trauma Acute Care Surg. 2018 May;84(5):819-825. doi: 10.1097/TA.0000000000001826. PMID 29432381
- [Background] Joint Committee to Create a National Policy to Enhance Survivability from Mass Casualty Shooting Events; Jacobs LM, Eastman A, Mcswain N, Butler FK, Rotondo M, Sinclair J, Wade DS, Fabbri WR. Improving Survival from Active Shooter Events: The Hartford Consensus. Bull Am Coll Surg. 2015 Sep;100(1 Suppl):32-4. No abstract available. PMID 26477133
- [Background] Eastridge BJ, Mabry RL, Seguin P, Cantrell J, Tops T, Uribe P, Mallett O, Zubko T, Oetjen-Gerdes L, Rasmussen TE, Butler FK, Kotwal RS, Holcomb JB, Wade C, Champion H, Lawnick M, Moores L, Blackbourne LH. Death on the battlefield (2001-2011): implications for the future of combat casualty care. J Trauma Acute Care Surg. 2012 Dec;73(6 Suppl 5):S431-7. doi: 10.1097/TA.0b013e3182755dcc. PMID 23192066
- [Background] Kotwal RS, Montgomery HR, Kotwal BM, Champion HR, Butler FK Jr, Mabry RL, Cain JS, Blackbourne LH, Mechler KK, Holcomb JB. Eliminating preventable death on the battlefield. Arch Surg. 2011 Dec;146(12):1350-8. doi: 10.1001/archsurg.2011.213. Epub 2011 Aug 15. PMID 21844425
- [Background] Biddinger PD, Baggish A, Harrington L, d'Hemecourt P, Hooley J, Jones J, Kue R, Troyanos C, Dyer KS. Be prepared--the Boston Marathon and mass-casualty events. N Engl J Med. 2013 May 23;368(21):1958-60. doi: 10.1056/NEJMp1305480. Epub 2013 May 1. No abstract available. PMID 23635020
- [Background] Teixeira PGR, Brown CVR, Emigh B, Long M, Foreman M, Eastridge B, Gale S, Truitt MS, Dissanaike S, Duane T, Holcomb J, Eastman A, Regner J; Texas Tourniquet Study Group. Civilian Prehospital Tourniquet Use Is Associated with Improved Survival in Patients with Peripheral Vascular Injury. J Am Coll Surg. 2018 May;226(5):769-776.e1. doi: 10.1016/j.jamcollsurg.2018.01.047. Epub 2018 Mar 29. PMID 29605726
- [Background] Scerbo MH, Holcomb JB, Taub E, Gates K, Love JD, Wade CE, Cotton BA. The trauma center is too late: Major limb trauma without a pre-hospital tourniquet has increased death from hemorrhagic shock. J Trauma Acute Care Surg. 2017 Dec;83(6):1165-1172. doi: 10.1097/TA.0000000000001666. PMID 29190257
- [Background] Scerbo MH, Mumm JP, Gates K, Love JD, Wade CE, Holcomb JB, Cotton BA. Safety and Appropriateness of Tourniquets in 105 Civilians. Prehosp Emerg Care. 2016 Nov-Dec;20(6):712-722. doi: 10.1080/10903127.2016.1182606. Epub 2016 May 31. PMID 27245978
- [Background] Beaucreux C, Vivien B, Miles E, Ausset S, Pasquier P. Application of tourniquet in civilian trauma: Systematic review of the literature. Anaesth Crit Care Pain Med. 2018 Dec;37(6):597-606. doi: 10.1016/j.accpm.2017.11.017. Epub 2018 Jan 5. PMID 29309952
- [Background] Butler FK Jr, Holcomb JB, Giebner SD, McSwain NE, Bagian J. Tactical combat casualty care 2007: evolving concepts and battlefield experience. Mil Med. 2007 Nov;172(11 Suppl):1-19. doi: 10.7205/milmed.172.supplement_1.1. PMID 18154234
- [Background] Jacobs LM, Burns KJ, Langer G, Kiewiet de Jonge C. The Hartford Consensus: A National Survey of the Public Regarding Bleeding Control. J Am Coll Surg. 2016 May;222(5):948-55. doi: 10.1016/j.jamcollsurg.2016.02.013. Epub 2016 Mar 31. No abstract available. PMID 27113518
- [Background] Sidwell RA, Spilman SK, Huntsman RS, Pelaez CA. Efficient Hemorrhage Control Skills Training for Healthcare Employees. J Am Coll Surg. 2018 Feb;226(2):160-164. doi: 10.1016/j.jamcollsurg.2017.11.003. Epub 2017 Nov 16. PMID 29155270
- [Derived] McCarty JC, Hashmi ZG, Herrera-Escobar JP, de Jager E, Chaudhary MA, Lipsitz SR, Jarman M, Caterson EJ, Goralnick E. Effectiveness of the American College of Surgeons Bleeding Control Basic Training Among Laypeople Applying Different Tourniquet Types: A Randomized Clinical Trial. JAMA Surg. 2019 Oct 1;154(10):923-929. doi: 10.1001/jamasurg.2019.2275. PMID 31339533

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-04-03): https://cdn.clinicaltrials.gov/large-docs/79/NCT03538379/Prot_SAP_000.pdf